CLINICAL TRIAL: NCT07161752
Title: Applied Forces During Neonatal Ventilation With Different Face Masks: a Randomized Crossover Manikin Study.
Brief Title: Applied Forces During Neonatal Ventilation With Different Face Masks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Professor, University of Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UNIPDNewborn25
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Face Mask Ventilation in Neonatal Resuscitation

STUDY DESIGN:
Intervention Model Description: Manikin study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anatomical face mask 1 (Experimental)
  Interventions: Device: Anatomical face mask 1
- Anatomical face mask 2 (Active Comparator)
  Interventions: Device: Anatomical face mask 2
- Round face mask (Active Comparator)
  Interventions: Device: Round face mask

INTERVENTIONS:
Device: Anatomical face mask 1 — Providing face mask ventilation in a neonatal manikin using a model of anatomical face mask
  Arms: Anatomical face mask 1
Device: Anatomical face mask 2 — Providing face mask ventilation in a neonatal manikin using another model of anatomical face mask
  Arms: Anatomical face mask 2
Device: Round face mask — Providing face mask ventilation in a neonatal manikin using a model of round face mask
  Arms: Round face mask

SUMMARY:
This trial compares the applied forces exerted on the face of a modified preterm neonatal manikin with three different face masks. Additionally, percentages of ventilation time with mask leak <25%, and participants' opinion about perceived applied forces, difficulty in achieving an effective ventilation, and difficulty in obtaining a good mask seal are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Level III neonatal intensive care unit (NICU) consultants, pediatric residents and anesthesiology residents

Exclusion Criteria:

* Refusal to participate

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Applied forces | 1 minute
  The force applied on the manikin head by the operator during the procedure

SECONDARY OUTCOMES:
Mask leak | 1 minute
  Mask leak (measured as percentage of ventilation time with leak less than 25% around the mask)
Participant opinion | 2 minutes
  Participants' opinions on the face masks (assessed using a Likert scale, from 1 lowest grade to 5 highest grade)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Università di Padova, Padua, Italy

REFERENCES:
- [Background] Cavallin F, Zamunaro A, Maglio S, Villani PE, Bua B, Gallo D, Menciassi A, Tognarelli S, Trevisanuto D. Applied forces with partially vs. fully inflated face masks during neonatal ventilation: a randomized crossover manikin trial. Pediatr Res. 2025 Aug 27. doi: 10.1038/s41390-025-04308-2. Online ahead of print. PMID 40866603
- [Background] Cavallin F, Sala C, Maglio S, Bua B, Villani PE, Menciassi A, Tognarelli S, Trevisanuto D. Applied forces with direct versus indirect laryngoscopy in neonatal intubation: a randomized crossover mannequin study. Can J Anaesth. 2023 May;70(5):861-868. doi: 10.1007/s12630-023-02402-9. Epub 2023 Feb 14. PMID 36788198
- [Background] Gordon JK, Bertram VE, Cavallin F, Parotto M, Cooper RM. Direct versus indirect laryngoscopy using a Macintosh video laryngoscope: a mannequin study comparing applied forces. Can J Anaesth. 2020 May;67(5):515-520. doi: 10.1007/s12630-020-01583-x. Epub 2020 Mar 9. PMID 32152886